CLINICAL TRIAL: NCT04580706
Title: The Effect of Frailty and Other Geriatric Syndromes on the Prognosis of Elderly Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Sun Ying, Director of department geriatrics, Beijing Friendship Hospital, Beijing Friendship Hospital
Other Study IDs: 2020-P2-097-01
Record Dates: First submitted 2020-09-11; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: ACS; Frail Elderly Syndrome; Elderly Patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: this is an observational study with none intervention — this is an observational study with none intervention

SUMMARY:
This is a prospective observational clinical trail which will recruit 1000-1500 participants over 65 years with frailty and acute coronary syndrome (ACS) in Beijing Friendship hospital. The investigators will conduct frailty assessment (FRAIL scale, CFS, SPPB), comorbidities, functional status (Barthel index, ADL, IADL), nutritional risk (MNA-SF), and then observe the clinical outcomes of elderly ACS participants with frailty. Then, the investigators will follow-up these participants separately in 1,3,6 and 12months, the anticipate follow-up time is 1 year. According to the follow-up results, investigators will evaluate the impact of frailty and other senile syndromes on the short-term and long-term prognosis of ACS, and develop a scoring system for the prognosis evaluation of elderly ACS participants.

ELIGIBILITY:
Inclusion Criteria:

* Elderly participants over 65
* Clinical diagnosis of acute coronary syndrome
* Must be able to follow-up
* Sign in the informed consent

Exclusion Criteria:

* Myocardial infarction caused by other acute disease
* Mental disorders who cannot cooperate to complete the assessment
* Severe liver dysfunction, kidney disease (CKD 5), end-stage malignant tumor
* Totally disabled and bedridden

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This registry will include consecutive patients age ≥65 years admitted for ACS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Death | During hospitalization, assessed up to 2 months
  All-cause death and cardiac death events
Major Adverse Cardiac and Cerebrovascular events | During hospitalization, assessed up to 2 months
  Major Adverse Cardiac and Cerebrovascular events including heart failure, cardiac shock, malignant arrhythmia, myocardial infarction, revascularization, and cerebral infarction
Death | 1 year
  All-cause death and cardiac death events
Major Adverse Cardiac and Cerebrovascular events | 1 year
  Major Adverse Cardiac and Cerebrovascular events including heart failure, cardiac shock, malignant arrhythmia, myocardial infarction, revascularization, and cerebral infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship hospital, Beijing, Beijing Municipality, China